CLINICAL TRIAL: NCT03479619
Title: Comparison of Three Lancing Devices Regarding Capillary Blood Volume and Lancing Pain Intensity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HTL-Strefa S.A. (Industry)
Collaborators: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 010617
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: lancing device; lancet
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- A/28/1 (Experimental): Lancing device A with personal lancet of size 28 G and minimum puncture depth.
  Interventions: Device: Lancing device A; Device: 28 G lancet; Other: Lancing depth setting (1)
- A/28/5 (Experimental): Lancing device A with personal lancet of size 28 G and maximum puncture depth.
  Interventions: Device: Lancing device A; Device: 28 G lancet; Other: Lancing depth setting (5)
- A/30/1 (Experimental): Lancing device A with personal lancet of size 30 G and minimum puncture depth.
  Interventions: Device: Lancing device A; Device: 30 G lancet; Other: Lancing depth setting (1)
- A/30/5 (Experimental): Lancing device A with personal lancet of size 30 G and maximum puncture depth.
  Interventions: Device: Lancing device A; Device: 30 G lancet; Other: Lancing depth setting (5)
- A/33/1 (Experimental): Lancing device A with personal lancet of size 33 G and minimum puncture depth.
  Interventions: Device: Lancing device A; Device: 33 G lancet; Other: Lancing depth setting (1)
- A/33/5 (Experimental): Lancing device A with personal lancet of size 33 G and maximum puncture depth.
  Interventions: Device: Lancing device A; Device: 33 G lancet; Other: Lancing depth setting (5)
- B/28/1 (Experimental): Lancing device B with personal lancet of size 28 G and minimum puncture depth.
  Interventions: Device: Lancing device B; Device: 28 G lancet; Other: Lancing depth setting (1)
- B/28/5 (Experimental): Lancing device B with personal lancet of size 28 G and maximum puncture depth.
  Interventions: Device: Lancing device B; Device: 28 G lancet; Other: Lancing depth setting (5)
- B/30/1 (Experimental): Lancing device B with personal lancet of size 30 G and minimum puncture depth.
  Interventions: Device: Lancing device B; Device: 30 G lancet; Other: Lancing depth setting (1)
- B/30/5 (Experimental): Lancing device B with personal lancet of size 30 G and maximum puncture depth.
  Interventions: Device: Lancing device B; Device: 30 G lancet; Other: Lancing depth setting (5)
- B/33/1 (Experimental): Lancing device B with personal lancet of size 33 G and minimum puncture depth.
  Interventions: Device: Lancing device B; Device: 33 G lancet; Other: Lancing depth setting (1)
- B/33/5 (Experimental): Lancing device B with personal lancet of size 33 G and maximum puncture depth.
  Interventions: Device: Lancing device B; Device: 33 G lancet; Other: Lancing depth setting (5)
- C/28/1 (Experimental): Lancing device C with personal lancet of size 28 G and minimum puncture depth.
  Interventions: Device: Lancing device C; Device: 28 G lancet; Other: Lancing depth setting (1)
- C/28/5 (Experimental): Lancing device C with personal lancet of size 28 G and maximum puncture depth.
  Interventions: Device: Lancing device C; Device: 28 G lancet; Other: Lancing depth setting (5)
- C/30/1 (Experimental): Lancing device C with personal lancet of size 30 G and minimum puncture depth.
  Interventions: Device: Lancing device C; Device: 30 G lancet; Other: Lancing depth setting (1)
- C/30/5 (Experimental): Lancing device C with personal lancet of size 30 G and maximum puncture depth.
  Interventions: Device: Lancing device C; Device: 30 G lancet; Other: Lancing depth setting (5)
- C/33/1 (Experimental): Lancing device C with personal lancet of size 33 G and minimum puncture depth.
  Interventions: Device: Lancing device C; Device: 33 G lancet; Other: Lancing depth setting (1)
- C/33/5 (Experimental): Lancing device C with personal lancet of size 33 G and maximum puncture depth.
  Interventions: Device: Lancing device C; Device: 33 G lancet; Other: Lancing depth setting (5)

INTERVENTIONS:
Device: Lancing device A — Glucoject Dual Plus lancing device
  Arms: A/28/1; A/28/5; A/30/1; A/30/5; A/33/1; A/33/5
Device: Lancing device B — Droplet lancing device
  Arms: B/28/1; B/28/5; B/30/1; B/30/5; B/33/1; B/33/5
Device: Lancing device C — Commercially available lancing device
  Arms: C/28/1; C/28/5; C/30/1; C/30/5; C/33/1; C/33/5
Device: 28 G lancet — Droplet 28 G
  Arms: A/28/1; A/28/5; B/28/1; B/28/5; C/28/1; C/28/5
Device: 30 G lancet — Droplet personal lancet 30 G
  Arms: A/30/1; A/30/5; B/30/1; B/30/5; C/30/1; C/30/5
Device: 33 G lancet — Droplet personal lancet 33 G
  Arms: A/33/1; A/33/5; B/33/1; B/33/5; C/33/1; C/33/5
Other: Lancing depth setting (1) — The lowest depth setting (1)
  Arms: A/28/1; A/30/1; A/33/1; B/28/1; B/30/1; B/33/1; C/28/1; C/30/1; C/33/1
Other: Lancing depth setting (5) — The highest depth setting (5)
  Arms: A/28/5; A/30/5; A/33/5; B/28/5; B/30/5; B/33/5; C/28/5; C/30/5; C/33/5

SUMMARY:
A randomized single-blind study with the use of three lancing devices equipped with personal lancets. Every device will be studied for three lancet sizes: 28G, 30G, and 33G with the minimum and maximum puncture depth setting.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosed diabetes type 1 or 2 ,
* aged 18 - 50,
* period of suffering from diabetes >2 years,
* performing on average 3-8 daily measurements of glycaemia,
* glycaemia at the moment of the beginning of the study between 70 and 200 mg/dl.

Exclusion Criteria:

* glycaemia below 70 mg/dl or glycaemia above 200 mg/dl at the moment of the beginning of the study,
* previously diagnosed hemorrhagic diathesis or heavy bleedings in the past (also those without a medical diagnosis),
* anticoagulant (thrombolytic medication) therapy within 3 weeks prior to the study or on the day of the study,
* non steroidal anti-inflammatory drugs (NSAID) treatment 1 week prior to the study or on the day of the study,
* patients with signs of dehydration,
* patients who are currently participating in another clinical study,
* currently diagnosed or reported by the patient skin diseases, nervous system diseases, psychiatric diseases, etc., which, in the opinion of the person conducting the study, disqualify the patient from the participation in the study, in care for the patient's well-being.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Volume (uL) of blood in the capillary tube | 1 - 3.5 hours (on average 2.5 hours) plus observation time after study 30 min
  Examination of the volume of blood obtained after puncturing a fingertip with the use of 3 lancing devices set to minimum and maximum puncture depth, with the use of various-sized personal lancets (28G, 30G, and 33G).
  The volume of blood sample will be measured with the use of capillary tubes calibrated for the volume of 10 μl and a graduated ruler.

SECONDARY OUTCOMES:
The intensity of pain perceived by the patient assessed with the use of the VAS (Visual Analog Scale). | 1 - 3.5 hours (on average 2.5 hours) plus observation time after study 30 min
  Examination of the intensity of pain perceived when puncturing a fingertip with the use of 3 lancing devices set to minimum and maximum puncture depth, with the use of various-sized personal lancets (28G, 30G, and 33G).

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Szadkowska, PhD,Md, Principal Investigator — Medical University of Lodz
Locations (1):
- Nzoz Magmed, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mianowska B, Mlynarski W, Szadkowska I, Szadkowska A. Evaluation of Three Lancing Devices: What Do Blood Volume and Lancing Pain Depend On? J Diabetes Sci Technol. 2021 Sep;15(5):1076-1083. doi: 10.1177/1932296820949930. Epub 2020 Aug 17. PMID 32856497